CLINICAL TRIAL: NCT06244836
Title: Comparison of Two Postoperative Infection Prevention Bundles in Colorectal Surgery. A Pragmatic Multicenter Cohort Study.
Brief Title: Comparison of Two Bundles of Care to Reduce Surgical Site Infection in Colorectal Surgery (CCR-VINCat 2)
Acronym: CCR-VINCat2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Granollers (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CCR-VINCat2
Record Dates: First submitted 2024-01-15; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Colon Cancer; Rectal Cancer; Surgical Site Infection
Keywords: Surveillance; Surgical site infection; Colorectal surgery; Prevention; Preventive measures; Bundle of care
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: The study compare three phases: a baseline period before bundle implementation (Baseline Group), from January 2011 to June 2016; a Bundle-1 period after the implementation of a six-measure bundle (Bundle-1 Group), from July 2016 to June 2018; and a Bundle-2 period after the implementation of a ten-measure bundle (Bundle-2 Group), from July 2018 to December 2022
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline group (No Intervention): Patients included in the Catalan Nosocomial Infection surveillance Program (VINCat) program, and operated on colorectal surgery before bundle implementation, from January 2011 to June 2016
- Implementation of a six-measures Bundle-1 (Bundle 1 Group) (Experimental): Bundle-1 period after the implementation of a six-measure bundle, from July 2016 to June 2018
  Interventions: Other: Implementation of a bundle of care
- Implementation of a ten-measures Bundle-2 (Bundle 2 Group) (Experimental): Bundle-2 period after the implementation of a ten-measure bundle, from July 2018 to December 2022
  Interventions: Other: Implementation of a bundle of care

INTERVENTIONS:
Other: Implementation of a bundle of care
  Arms: Implementation of a six-measures Bundle-1 (Bundle 1 Group); Implementation of a ten-measures Bundle-2 (Bundle 2 Group)

SUMMARY:
There is controversy about the maximum number of elements to be included in a surgical site infection (SSI) prevention bundle and the possibility of its implementation at a multi-center level.

This study analyzes SSI rates in colorectal surgery after the implementation of two preventive bundles.

The investigators hypothesized that the thorough introduction of a well-designed large bundle of best practice preventive measures would result in good adherence and greater reduction of SSI rates after colorectal surgery.

DETAILED DESCRIPTION:
To better understand the impact of adding new measures to an established bundle within a national surveillance program and to measure the effectiveness of each specific measures, the effect of a six-measure and a ten-measure bundle sequentially implemented on a large series of elective colorectal procedures from 2011 to 2022 was analized. In addition, it will be investigated whether taking advantage of a national surveillance programme for post-operative infections can facilitate the implementation of the packages.

Setting and patients. This is a pragmatic, cohort, multicentre study of a network of 65 public and private hospitals prospectively collecting data from elective colorectal surgery to minimise surgical site infection (SSI) rates and improve care. Prospective surveillance is conducted by each hospital's infection control team to ensure adequate data collection with a mandatory minimum follow-up of 30 days after surgery and electronic chart review checking readmissions, emergency department visits, microbiological and radiological data.

Patients undergoing elective colorectal surgery between January 2011 and December 2022 will be included. Cases with class 2 (clean-contaminated) and 3 (contaminated) wounds, according to the National Healthcare Safety Network classification, will be followed up. Patients with class 4 wounds (peritonitis) and previous ostomies are excluded.

Three sequential phases will be compared: a baseline period before package implementation (Baseline Group), from January 2011 to June 2016; a Bundle-1 period after implementation of a package of six measures (Bundle-1 Group), from July 2016 to June 2018; and a Bundle-2 period after implementation of a package of ten measures (Bundle-2 Group), from July 2018 to December 2022.

Definitions, study results and variables. The SSIs are defined according to the definitions of the Centers for Disease Control and Prevention.

The primary objective will be to analyse the effect of the implementation of the package on the prevention of SSIs and their subtypes and to assess compliance and effectiveness of individual measures. Secondary outcomes will be length of stay, mortality and micro-organisms causing SSIs.

Intervention. In the Reference Group, some measures such as intravenous antibiotic prophylaxis and the use of laparoscopy were included as standard clinical practice. In Bundle-1, six well-documented colorectal-specific measures were introduced: intravenous antibiotic prophylaxis, laparoscopy, oral antibiotic prophylaxis, mechanical bowel preparation, normothermia and double-ring plastic wound retractor. In Bundle-2, four additional general measures were incorporated in addition to the above: adequate depilation, skin antisepsis with 2% chlorhexidine gluconate in alcohol, perioperative glucose control and instrument change before wound closure.

ELIGIBILITY:
Inclusion Criteria:

* Colon or rectal elective surgery.

Exclusion Criteria:

Peritonitis at the time of intervention ("dirty" surgery) Patients who underwent multiple procedures during the same surgery, for example resection of liver metastases Centers that performed less tan 10 surgical procedures annually Centers that have not been able to ensure prospective surveillance during hospitalization or effective monitoring of cases within 30 days of the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32205 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Surgical site infection (SSI) incidence within 30 days of surgery according to the Centers for Disease Control and Prevention (CDC) criteria. | 30 days
  Overall surgical site infection (SSI) rate will be defined as any infection originating in surgical wounds or the organs/spaces opened or manipulated during an operative procedure. The incidence of SSI will be measured as events per 100 procedures included.

SECONDARY OUTCOMES:
Organ/space surgical infection rate within 30 days of surgery according to the Centers for Disease Control and Prevention (CDC) criteria. | 30 days
  Specific organ/space surgical infection (O/S-SSI) rate. O/S-SSI is the infection that involves any part of the anatomy in organs and spaces other than the incision, which is opened or manipulated during operation. he incidence of O/S-SSI will be measured as events per 100 procedures included.
Hospital type-Surgical infection rate within 30 days of surgery according to the Centers for Disease Control and Prevention (CDC) criteria. | 30 days
  Comparison of SSIs rates among the three hospitals groups, according to their size. The hospitals are classified into three groups according to their complexity and number of hospital beds: >500 beds; 200-500 beds; ≤200 beds.

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Badia, MD, PhD, Principal Investigator — Hospital General de Granollers
Locations (1):
- Hospital General de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be shared if requested